CLINICAL TRIAL: NCT01329588
Title: Periodical Presumptive Treatment of Gonorrhoea in Female Sex Workers: Impact on Prevalence of the Disease in Sex Workers and Their Clients
Brief Title: Periodical Presumptive Treatment for the Control of Gonococcal Infections Among Sex Workers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Ministry of Health, Benin (Other Government)
Responsible Party: Michel Alary, Unité de recherche en santé des populations
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR-002-947
Record Dates: First submitted 2011-02-14; First posted 2011-04-06 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Neisseria Gonorrhoeae Infection; Chlamydia Trachomatis; HIV
Keywords: Female sex workers; West Africa; Presumptive treatment; Sexually transmitted infections
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases | interventions — Azithromycin; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Monthly placebo
- Treatment arm (Experimental)
  Interventions: Drug: Monthly antibiotic

INTERVENTIONS:
Drug: Monthly antibiotic — Azithromycin 1g per os once at months 1, 4 and 7 Ciprofloxacin 500 mg per os once at months 2, 3, 5, 6, 8 and 9
  Other Names: Zithromax and cipro
  Arms: Treatment arm
Drug: Monthly placebo — Azithromycin placebo (sugar pill) per os once at months 1, 4 and 7 Ciprofloxacin placebo (sugar pill) per os once at months 2, 3, 5, 6, 8 and 9
  Arms: Sugar pill

SUMMARY:
In the early years of the HIV epidemic in Africa, female sex workers (FSWs) were identified as a high-prevalence, high-incidence, core group among whom the extraordinary prevalence of other sexually transmitted infections (STIs) facilitated transmission of the virus to their clients, who then infected low-risk women not involved in the sex trade. In resource-poor settings, control of Neisseria gonorrhoeae (NG) and Chlamydia trachomatis (CT) among FSWs is difficult. The purpose of this study is to determine whether periodical antibiotic treatment (PAT) is effective in controlling these infections among West African FSWs.

The study is designed as a cluster-randomized double-blind placebo-controlled trial conducted in West Africa. The study population consists of "seaters" FSWs who work from their homes in well-defined areas. Clusters will be paired according to their size and demographic characteristics of FSWs and clients. Within each pair, one cluster will be randomly allocated to the intervention and the other to the placebo group.

At enrollment, participants will be interviewed, a pelvic examination performed, cervical swabs obtained for NG and CT polymerase chain reaction (PCR), and current cervicitis or vaginitis managed syndromically. Blood specimens will be obtained for HIV testing. All participants will be given free condoms and counseled on risk reduction.

Monthly follow-up will be conducted within FSW communities, alternating with clinic visits where cervical samples will be collected. Study drugs (azithromycin 1 g and ciprofloxacin 500 mg, and their identical placebos) will be distributed every month according to a predefined schedule: directly-observed intake of azithromycin at months 1, 4 and 7, and ciprofloxacin at months 2, 3, 5, 6, 8 and 9.

Data will be analyzed with SAS. The investigators will assess the time trends in NG and CT prevalence separately in both study groups using χ2-for-trend.

DETAILED DESCRIPTION:
"Seaters" are older, more stable, better organized, and have a much higher prevalence of HIV infection than FSWs who roam the streets or part-time sex workers. These communities (from 3 to 114 FSWs per site) will be aggregated into 18 clusters (one cluster was composed of 1-10 FSW communities) based on geographical proximity. Over a one-year period, FSWs from these clusters presenting to dedicated clinics will be invited to participate. In addition, field workers will visit FSWs at home or at prostitution sites to provide information about the trial and seek participation.

Clusters will be paired according to their size and demographic characteristics of FSWs and clients. Within each pair, one cluster will be randomly allocated to the intervention and the other to the placebo group using pre-coded envelopes. With an average of 35 FSWs per cluster, the required number of cluster pairs is estimated at 8.7 to detect a 50% reduction in NG prevalence, assuming a baseline prevalence of 25%, 80% power and 5% alpha error.

ELIGIBILITY:
Inclusion Criteria:

* Female sex worker (seater) from one of the selected clusters

Exclusion Criteria:

* Allergy to study drugs
* Pregnancy
* Intention to leave the city within the next 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2001-03; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Presence of gonococcal infection | 3 months
  Cervical samples for NG PCR will be collected at the clinic visit planned at months 3 (between 45-134 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.
Presence of gonococcal infection | 6 months
  Cervical samples for NG PCR will be collected at the clinic visit planned at months 6 (between 135-224 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.
Presence of gonococcal infection | 9 months
  Cervical samples for NG PCR will be collected at the clinic visit planned at months 9 (between 225-315 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.

SECONDARY OUTCOMES:
Presence of chlamydia infection | 3 months
  Cervical samples for CT PCR will be collected at the clinic visit planned at months 3 (between 45-134 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.
Presence of chlamydia infection | 6 months
  Cervical samples for CT PCR will be collected at the clinic visit planned at months 6 (between 135-224 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.
Presence of chlamydia infection | 9 months
  Cervical samples for CT PCR will be collected at the clinic visit planned at months 9 (between 225-315 days after enrolment). Time trend in gonorrhoea prevalence will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Alary, MD, PhD, Principal Investigator — Centre de recherche, Centre hospitalier affilié universitaire de Québec
Locations (1):
- Dispensaire des infections sexuellement transmissibles, Cotonou, Benin

REFERENCES:
- [Derived] Labbe AC, Pepin J, Khonde N, Dzokoto A, Meda H, Asamoah-Adu C, Mayaud P, Mabey D, Demers E, Alary M. Periodical antibiotic treatment for the control of gonococcal and chlamydial infections among sex workers in Benin and Ghana: a cluster-randomized placebo-controlled trial. Sex Transm Dis. 2012 Apr;39(4):253-9. doi: 10.1097/OLQ.0b013e318244aaa0. PMID 22421690